CLINICAL TRIAL: NCT06385457
Title: The Effects of Mindhelper.dk: a Self-guided Digital Mental Health Promotion Service Targeting Young People
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry); Danske Regioner (Other); Jascha Fonden (Other); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Anna Paldam Folker, Head of Research, Professor, ph.d., University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24-2933
Record Dates: First submitted 2024-04-15; First posted 2024-04-26 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Mental Health Issue; Well-Being; Adolescents; Young Adults; Online Intervention; Internet-Based Intervention; Randomized Controlled Trial; Body Dissatisfaction
Keywords: Self-guided; Prevention; Well-being; eHealth; Promotion; Adolescents; Young adults; Body Appreciation

STUDY DESIGN:
Intervention Model Description: Participants will be recruited via social media, and randomly allocated to an intervention group (receiving information about Mindhelper.dk) or a control group (no information about Mindhelper.dk). Outcomes, will be measured at 2-, 6-, and 12-weeks post-randomization and analysed using the intention-to-treat approach.
  According to the investigators' power calculation, at least 3,142 participants (1,571 in each group) are required at follow-up 2 weeks after the randomization (primary endpoint). In the test phase, the investigators retrieved a response proportion of 64% for this follow-up survey. Assuming a similar retention proportion the investigators aim to include 4910 participants at baseline. The proportion of participants responding to the follow-up surveys will be regularly reviewed to evaluate if the assumption on retention is correct or if the number of participants included should be increased or decreased.
Who Masked: Investigator
Masking Description: The participants are partly masked. The control group will be masked; however, the intervention group will not be masked.
  There is no care provider nor outcome assessor as all measures are self-reported and collected through online questionnaires.
  Analyses of data and interpretation of results will be done masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive information about Mindhelper.dk and inspiration on how to use Mindhelper through text-messages during the study period.
  Interventions: Behavioral: Mindhelper- A national youth mental health promotion website
- Control group (No Intervention): The control group does not receive information about Mindhelper.dk, until after completion of the last follow-up questionnaire.

INTERVENTIONS:
Behavioral: Mindhelper- A national youth mental health promotion website — Mindhelper is an open-access, digital self-directed mental health service that provides information, self-help tools and guidance to young people in Denmark.
  Arms: Intervention group

SUMMARY:
In a two-armed randomized controlled trial 15-25-year-olds will be recruited via social media to evaluate the effectiveness of Mindhelper.dk; a Danish self-guided, digital, mental health service offering information, self-help tools, and guidance to young people. Participants will be randomly allocated to an intervention group (receiving information about Mindhelper.dk) or a control group (no information about Mindhelper.dk). Outcomes, including well-being (WHO5), psychological functioning (SWEMWBS), help-seeking intentions, and body appreciation (2-item BAS-2SF), will be measured at 2-, 6-, and 12-weeks post-randomization and analyzed using the intention-to-treat approach. Qualitative interviews with intervention group participants will provide complementary insights, and a cost-effectiveness analysis will also be conducted.

DETAILED DESCRIPTION:
A study protocol will be made publicly accessible upon acceptance for publication in a suitable journal

ELIGIBILITY:
-Aged 15-25

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Men, women, and others
Enrollment: 4910 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
General well-being measure by "The Well-Being Index WHO-5" (WHO5) | Baseline and randomization(T1), 2 weeks (T2), 6 weeks(T3) and 12 weeks (T4) after randomization.
  The WHO5 scores range between 0 and 100. The higher score, the higher level of well-being.
  The effects of Mindhelper on well-being are measured through surveys disseminated to the study participants. The primary assessment of effect is conducted at T2.

SECONDARY OUTCOMES:
Psychological functioning, measure by "The Short Warwick-Edinburgh Mental Well-Being Scale" (SWEMWBS). | Baseline and randomization(T1), 2 weeks (T2), 6 weeks(T3) and 12 weeks (T4) after randomization.
  The SWEMWBS scores range from 7 to 35, and higher scores indicate higher levels of mental wellbeing.
  The effects of Mindhelper on psychological functioning are measured through surveys disseminated to the study participants. The primary assessment of effect is conducted at T2.

OTHER OUTCOMES:
Intentions of help-seeking | Baseline and randomization(T1), 6 weeks(T3) and 12 weeks (T4) after randomization.
  As the investigators have developed the questions used to assess intentions of help-seeking no validated ranging of score exists.
  The effects of Mindhelper on intentions to help-seeking are measured through surveys disseminated to the study participants. The primary assessment of effect is conduct at T3.
Body Appreciation measured by the "2-items Short forms of the Body Appreciation Scale-2" (2-item BAS-2SF). | Baseline and randomization(T1), 2 weeks (T2), 6 weeks(T3) and 12 weeks (T4) after randomization.
  The BAS-2SF uses a 5-point Likert scale for responses, ranging from 1 (Never) to 5 (Always), thus for 2-item BAS-2SF the score ranges from 2 to 10. Higher scores indicate greater body appreciation.
  The effects of Mindhelper on body appreciation are measured through surveys disseminated to the study participants. The primary assessment of effect is conduct at T2.

CONTACTS AND LOCATIONS:
Overall Officials: Anna P Folker, Principal Investigator — National Institute of Public Health, University of Southern Denmark
Locations (1):
- National Institute of Public Health (NIPH), University of Southern Denmark, Copenhagen, Copenhagen K, Denmark

IPD SHARING:
Plan to Share IPD: Yes
It will be possible to share IPD, but no plans of this have yet been made.
Supporting Information: Study Protocol, SAP
Time Frame: Before end of data collection
Access Criteria: Will be published in open repositories

REFERENCES:
- [Background] Hoffmann SH, Paldam Folker A, Buskbjerg M, Paldam Folker M, Huber Jezek A, Lyngso Svarta D, Nielsen Solvhoj I, Thygesen L. Potential of Online Recruitment Among 15-25-Year Olds: Feasibility Randomized Controlled Trial. JMIR Form Res. 2022 May 25;6(5):e35874. doi: 10.2196/35874. PMID 35612877
- [Derived] Hoffmann SH, Kusier AO, Mairey IP, Folker AP, Thygesen LC. A Self-Guided Digital Mental Health Promotion Service Targeting Young People: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 10;14:e73736. doi: 10.2196/73736. PMID 40929726